CLINICAL TRIAL: NCT00382811
Title: Multi-Center, Randomized, Double-Blind, Phase III Efficacy Study Comparing Phenoxodiol in Combination With Carboplatin Versus Carboplatin With Placebo in Patients With Platinum-Resistant or Platinum-Refractory Late-Stage Epithelial Ovarian, Fallopian or Primary Peritoneal Cancer Following at Least Second Line Platinum Therapy
Brief Title: OVATURE (OVArian TUmor REsponse) A Phase III Study of Weekly Carboplatin With and Without Phenoxodiol in Patients With Platinum-Resistant, Recurrent Epithelial Ovarian Cancer
Acronym: OVATURE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MEI Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NV06-0039
Record Dates: First submitted 2006-09-28; First posted 2006-10-02 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Fallopian Tube Cancer; Peritoneal Neoplasms; Ovarian Cancer
Keywords: Recurrent Ovarian Epithelial Cancer; Stage IV Ovarian Epithelial Cancer; Peritoneal Cavity Cancer; Stage III Ovarian Epithelial Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Peritoneal Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — phenoxodiol; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): Daily Phenoxodiol + weekly carboplatin
  Interventions: Drug: phenoxodiol; Drug: carboplatin
- 2 (Active Comparator): Daily phenoxodiol placebo + weekly carboplatin
  Interventions: Drug: carboplatin; Drug: placebo

INTERVENTIONS:
Drug: phenoxodiol — 400mg phenoxodiol three times daily in 28 day cycles.
  Arms: 1
Drug: carboplatin — AUC=2 weekly in 28 day cycles
Drug: placebo — every 8 hours daily in 28 day cycles
  Arms: 2

SUMMARY:
The purpose of this project is to see if weekly carboplatin compared with phenoxodiol in combination with weekly carboplatin, is effective against late stage ovarian cancer and to see what, if any, side-effects of treatment may result.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed ovarian, fallopian, or primary peritoneal carcinoma of epithelial origin
* Recurrent or persistent advanced disease
* Have measurable disease
* Undergone at least two courses of therapy with a platinum drug (cisplatin or carboplatin) and have responded to the first of those courses of therapy as determined by either Response Evaluation Criteria in Solid Tumors (RECIST) or Gynecologic Cancer Intergroup (GCIG) criteria
* Disease relapse as determined by either RECIST or GCIG criteria within 6 months of completion of the second or greater course of platinum therapy using a 2-, 3- or 4-weekly regimen and platinum-free interval of no greater than 6 months at the time of enrollment, being the time taken from the last day of platinum therapy
* Any number of previous courses of platinum therapy or non-platinum therapy
* Likely to survive at least 3 months
* Karnofsky performance score of at least 60%
* Have adequate physiological function without evidence of major organ dysfunction as evidenced by:

  * serum creatinine < 1.5 mg/dl
  * serum transaminase levels ≤ 3 x the upper limit of normal (ULN) for the reference laboratory and
  * bilirubin level < ULN
* Have adequate hematological function defined by:

  * platelets > 100,000/mm3
  * white cell counts (WCC) > 3,000/mm3
  * neutrophils > 1,500/mm3
  * hemoglobin > 8.0 g/dl
* Aged > 18
* Be able to understand the risks and benefits of the study and give written informed consent to participation.

Exclusion Criteria:

* Patients with mucinous histological type of ovarian cancer
* Patients who have failed to show a clinical response (RECIST or GCIG criteria) to at least one prior course of platinum therapy
* Patients with active infection
* Patients with concurrent severe and/or uncontrolled medical disease (e.g., uncontrolled diabetes, hypertension, ischemic heart disease, congestive heart failure, etc.)
* Patients with a history of chronic active hepatitis or cirrhosis
* Patients with HIV
* Patients with active central nervous system (CNS) metastases. Patients with known CNS metastases must have received prior radiation therapy, and CNS metastatic disease must be stable for 4 weeks.
* Patients who have not recovered from the acute effects of any prior anti-neoplastic therapy
* Patients with known hypersensitivity to platinum drugs that cannot be managed with concomitant medication.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2006-10; Primary Completion 2009-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The primary efficacy end-point is progression-free survival (PFS). PFS is the time from randomization until disease progression or death | Progression Free Survival

SECONDARY OUTCOMES:
The secondary efficacy end-point is overall survival (OS) | Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Daniel P Gold, PhD, Study Director — MEI Pharma, Inc.
Locations (70):
- United States (37):
  - Arizona Clinical Research Center, Inc., Tuscon, Arizona
  - Glendale Adventist, Glendale, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Gynecology Oncology Associates, Newport Beach, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Hematology Oncology, PC (Carl and Dorothy Bennett Cancer Center), Stamford, Connecticut
  - Gynecologic Oncology Associates, Pembroke Pines, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Medical College of Georgia Cancer Center, Augusta, Georgia
  - Associates in Women's Health, Wichita, Kansas
  - Hematology and Oncology Specialists, LLC, Metairie, Louisiana
  - Greater Baltimore Medical Centre, Baltimore, Maryland
  - Gynecologic Oncology of West Michigan, Grand Rapids, Michigan
  - Providence Hospital and Medical Centers, Southfield, Michigan
  - The Center for Cancer & Hematological Disease, Cherry Hill, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - The University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Schwartz Gynecologic Oncology, Brightwaters, New York
  - New York Downtown Hospital, New York, New York
  - University of Rochester Gynecologic Oncology Associates, Rochester, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Brody School of Medical at East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - OSU James Cancer Hospital & Solove Research Institute, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Chattanooga GYN Oncology, Chattanooga, Tennessee
  - Chattanooga's Program In Women's Oncology, Chattanooga, Tennessee
  - Hall and Martin MDS, P.C., Knoxville, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Hope Cancer Clinic, Brownsville, Texas
  - University of Texas Southwestern Medical Center Simmons Comprehensive Cancer Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Northern Virginia Pelvic Surgery Associates, Annadale, Virginia
  - Virginia Mason Medical Center Department of Hematology/Oncology, Seattle, Washington
- Australia (5):
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Mater Adult Hospital, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
- Belgium (2):
  - UZ Antwerpen, Edegem
  - UZ Leuven, Leuven
- Italy (2):
  - IEO- Istituto Europeo di Oncologia, Milan
  - Istitutio Fisioterapici Ospitaleri, Roma
- Poland (7):
  - Bialostockie Centrum Onkologii im. Marii Sklodowskiej-Curie Oddzial Onkologii Ginekologicznej, Bialystok
  - Ackademickie Centrum Kliniczne-Szpital, Akademii Medycznej w Gdansku, Gdansk
  - Centrum Onkologii-Instytut im. M. Sklodowskiej-Curie, Oddzial w Gliwicach, Gliwice
  - Centrum Onkologii - Instytut im. M. Sklodowskiej-Curie Oddzial w Krakowie Klinika Ginekologii Onkologicznej, Krakow
  - Centrum Onkologii Ziemi, Lublin
  - Ginekologiczno - Polozniczy Szpital Kliniczny AM im. K. Marcinkowskiego w Poznaniu SPZOZ Klinika Onkologii Ginekologicznej, Poznan
  - Centrum Onkologii-Instytut im. M. Sklodowskiej Curie Klinika Nowotworow Narzadow Plciowych Kobiecych, Warsaw
- Spain (6):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital General Universitario de Alicante, Alicante
  - Hospital General Vall d'Hebron, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital General Universitario de Valencia, Valencia
- United Kingdom (11):
  - Yeovil District Hospital, Yeovil, Somerset
  - Cancer Research UK Clinical Trials Unit Old Clinical Investigations Building, Birmingham
  - Ninewells Hospital, Dundee
  - Edinburgh Cancer Research Centre Western General Hospital, Edinburgh
  - The Beatson West of Scotland Cancer Centre, Glasgow
  - St James University Hospital, Leeds
  - Hammersmith Hospital, London
  - Cancer Research UK & UCL Cancer Trials Center, London
  - Clatterbridge Centre for Oncology, Metropolitan Borough of Wirral
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Royal Marsden NHS Foundation Trust, Sutton

REFERENCES:
- [Derived] Fotopoulou C, Vergote I, Mainwaring P, Bidzinski M, Vermorken JB, Ghamande SA, Harnett P, Del Prete SA, Green JA, Spaczynski M, Blagden S, Gore M, Ledermann J, Kaye S, Gabra H. Weekly AUC2 carboplatin in acquired platinum-resistant ovarian cancer with or without oral phenoxodiol, a sensitizer of platinum cytotoxicity: the phase III OVATURE multicenter randomized study. Ann Oncol. 2014 Jan;25(1):160-5. doi: 10.1093/annonc/mdt515. Epub 2013 Dec 5. PMID 24318743
- See also: Click here for more information on the study and sponsor. — http://www.marshalledwardsinc.com/